CLINICAL TRIAL: NCT06126523
Title: Effect of Extracorporeal Shock Wave Therapy Applied After Botulinum Toxin Injection on Ankle Plantar Flexor Spasticity in Stroke Patients: Placebo-controlled Double-blind Study.
Brief Title: Effect of ESWT Applied After Botulinum Toxin Injection on Ankle Spasticity in Stroke Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep Selimoğlu Ayneli, Lecturer PHD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSAYNELI
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Spasticity as Sequela of Stroke
Keywords: spasticity; ESWT; Botulinum Toxin
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT once (Active Comparator): A single session of rESWT will be applied on the same day after BTX-A injection.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy ONCE
- ESWT twice (Active Comparator): A total of 2 sessions of rESWT will be applied on the same day after BTX-A injection and on the 7th day after BTX-A.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy ONCE; Device: Radial Extracorporeal Shock Wave Therapy TWİCE
- Sham ESWT (Sham Comparator): A single session of placebo rESWT will be applied after BTX-A injection.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy SHAM

INTERVENTIONS:
Device: Radial Extracorporeal Shock Wave Therapy ONCE — rESWT application ONCE The points where rESWT will be applied will be determined under ultrasonography guidance. The pressure pulses will be focused on the injection site in the medial and lateral heads of the gastrocnemius muscle and the soleus muscle.
  Number of pulses: 1500 pulses Frequency: 6 Hz Energy level/Pressure: 2.2 bar air pressure Duration: 12 minutes
  Device to be used in research ELMED VIBROLITH ESWT SW. Give. 3.3 It is based on the principle that currents produced outside the body spread in the tissue in the form of sound waves.
  Arms: ESWT once; ESWT twice
Device: Radial Extracorporeal Shock Wave Therapy TWİCE — rESWT application TWİCE The points where rESWT will be applied will be determined under ultrasonography guidance. The pressure pulses will be focused on the injection site in the medial and lateral heads of the gastrocnemius muscle and the soleus muscle.
  A total of 2 sessions of rESWT will be applied on the same day after BTX-A injection and on the 7th day after BTX-A.
  Number of pulses: 1500 pulses Frequency: 6 Hz Energy level/Pressure: 2.2 bar air pressure Duration: 12 minutes
  Device to be used in research ELMED VIBROLITH ESWT SW. Give. 3.3 It is based on the principle that currents produced outside the body spread in the tissue in the form of sound waves.
  Arms: ESWT twice
Device: Radial Extracorporeal Shock Wave Therapy SHAM — Radial Extracorporeal Shock Wave Therapy- SHAM The points where rESWT will be applied will be determined under ultrasonography guidance. The pressure pulses will be focused on the injection site in the medial and lateral heads of the gastrocnemius muscle and the soleus muscle.
  Sham ESWT will be administered with the r-ESWT probe. The device will be switched on, the frequency, pressure and duration values will be set and then the device will be switched off and the probe will be kept in equal time with the active treatment, by playing a sound previously recorded during the real application.
  Arms: Sham ESWT

SUMMARY:
Stroke is the second most common cause of death and the third most important cause of disability worldwide, with an annual death rate of 5.5 million. Spasticity is a common condition in stroke patients and has a negative impact on daily living activities. BTX-A has been successfully used in the treatment of spasticity in patients with stroke. ESWT is a physical therapy method applying high intensity pressure waves.

ESWT has been increasingly used in the management of spasticity as a safe and effective method, but the literature about ESWT in spasticity is heterogeneous and the treatment protocols are not very clear about the number of applications.

The aim of this study is to determine the effects of rESWT treatment on ankle plantar flexors spasticity applied after BTX-A injection.

DETAILED DESCRIPTION:
In this double-blind randomized placebo-controlled trial, 45 patient (aged 18-75) diagnosed as stroke with appropriate criteria will be included.

Patients who meet the inclusion criteria for the study will be seperated into three groups with the randomizer.org randomization program.

Group I: A single session of rESWT will be applied on the same day after BTX-A injection.

Group II: A total of 2 sessions of rESWT will be applied on the same day after BTX-A injection and on the 7th day after BTX-A injection.

Group III: A single session of placebo rESWT will be applied after BTX-A injection.

BTX-A injections to gastrocnemius and soleus muscles will be performed under ultrasonography guidance. rESWT will be applied to the injection points in gastrocnemius and soleus muscles.

The pressure pulses will be focused on the injection site in the medial and lateral heads of the gastrocnemius muscle and the soleus muscle. (Number of pulses: 1500 pulses, frequency: 6 Hz, Energy level/Pressure: 2.2 bar air pressure, duration: 12 minutes) Patients will be evaluated by the same researcher before treatment, 2 weeks after treatment, 1 month after treatment and 3 months after treatment.

Patients will be evaluated using the Modified Ashworth Scale, Modified Tardieu Scale, Visual Analog Scale, 10 m walk test, Timed Up and Go Test, Timed Sit and Go Test, Barthel Activities of Daily Living Index, Functional Ambulation Scale, Brunnstrom Staging.

ELIGIBILITY:
Inclusion Criteria:

* Having an ischemic or hemorrhagic stroke, in subacute or chronic phase,
* Patients with ankle plantar flexor spasticity MAS score > 1 and patients who received BTX-A injection due to spasticity
* Stroke history of at least 3 months

Exclusion Criteria:

* History of neuromuscular disease
* Compared to the unaffected side; More than 50% reduction in dorsiflexion range of motion of the affected side
* Dynamic ankle contracture
* Affected side lower extremity surgery in the last 12 months
* Having Botox or phenol application to the affected gastrocnemius in the last 3 months
* Change in the dose of antispastic medication used in the last 3 months
* Infection/wound in the affected lower extremity
* Contraindications for ESWT (pregnancy, cancer, bleeding disorders, inflammatory disease, pacemakers or other electronic implants).
* Significant muscle atrophy or fibrosis of the target muscle (Heckmatt scale III and IV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-26 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient Evaluation Form | BEFORE TREATMENT
  Demographic information, stroke history, and medications used by all stroke patients included in the study will be recorded.
Modified Ashworth Scale (MAS) | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It is a method used to determine the severity of spasticity. It is based on the subjective rating of the resistance felt during the examination Modified Ashworth Scale is graded between 0 and 4 points. 0: No increase in muscle tone, 4: affected part is rigid in flexion or extension.
  It means that the higher the score the patient receives, the higher the degree of spasticity.
Modified Tardieu Scale (MTS) | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  The severity of muscle tone is evaluated at different determined speeds. The first angle at which an increase in resistance is detected in the joint is recorded. The range of motion is compared with the angle at completion.The minimum value in evaluating the joint angle is 0 degrees.The maximum value varies depending on the patient's joint.Higher angle value means worse result.
  Modified Tardieu Scale is rated between 0 and 5 points. 0: no resistance during passive motion, 5: The joint can not be moved. It means that the higher the score the patient receives, the higher the degree of spasticity.
10m walking test | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  Subjects are asked to walk at maximum speed in a 10-meter corridor. The time it takes them to complete the distance is measured in seconds with a stopwatch. The measurement is repeated three times and the average time of the three measurements is recorded.
Timed Up and Go Test | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  The person is asked to get up from the chair, walk 3 meters at a safe and normal pace, turn, walk back and sit on the chair, and the time is recorded in seconds.
Timed sit and stand test | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It is a test that evaluates the patient's sit-to-stand activity, lower extremity strength and dynamic balance. The number of times the patient sits and stands up within 30 seconds gives the test score.
Barthel Activities of Daily Living Index | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It is used to measure the independence of the individual in daily living activities.
Functional Ambulation Scale | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It classifies individuals between 0 and 5 according to the basic motor skills required for functional ambulation.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It is a scale used to measure contraction from a 10 cm horizontal axis.A score of zero means no contraction, and a score of ten means the most severe contraction felt.
  The higher the score the patient receives, the higher the degree of contraction.
Brunnstrom Staging | BEFORE TREATMENT, 2 WEEKS LATER AFTER TREATMENT, 1 MOUNTH LATER AFTER TREATMENT, 3MOUNTH LATER AFTER TREATMENT
  It classifies stroke patients with improvement in upper extremity, lower extremity and hand functions.

CONTACTS AND LOCATIONS:
Locations (1):
- SaglikBilimleriU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No